CLINICAL TRIAL: NCT02937909
Title: A Prospective Study With Historical Data Comparison to Evaluate the Benefits of Using a Range of Products From a Single Manufacturer for Training, Competencies in Wound Care and the Appropriate Use of Product
Brief Title: A Study to Evaluate the Benefits of Using a Range of Wound Care Products From a Single Manufacturer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Inadequate patient recruitment
Sponsor: BSN Medical Ltd. UK (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WMC 75/UK/15
Record Dates: First submitted 2016-08-31; First posted 2016-10-19 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Wound - in Medical Care
Keywords: woundcare community nursing competence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective Data (Experimental): Use of BSN medical UK range of wound dressings and compression products for 12 weeks treatment period Training and testing of woundcare nursing competencies Quality of Life questionnaire for patients
  Interventions: Other: Use of wound care products from a single manufacturer
- Historical data (No Intervention): Historical data from the three months prior to the study on time needed for nurse training, number of referrals to the Tissue Viability Team, costs of dressings used, number of patients with wounds treated, types of wounds, number of wound closures and duration of treatment .

INTERVENTIONS:
Other: Use of wound care products from a single manufacturer — The participating Healthcare Professionals will be asked to use BSN medical wound care products for the study duration
  Arms: Prospective Data

SUMMARY:
This study is designed to investigate whether the adoption of the use of a range of wound care products from a single manufacturer makes training in appropriate product selection more effective and results in more accurate selection of the appropriate product for the wound and for the patient's lifestyle, thereby incurring less waste and reducing the number of referrals by the community nursing team to the Tissue Viability Team.

One community nursing team will switch to using a full range of dressings and compression products from BSN medical UK for three months. Nurse training on the products will be given and nurse competencies and confidence in woundcare and appropriate product selection will be tested at the start and end of the study.

The number and type of referrals to the Tissue Viability Team will be measured.

Total anonymised data on numbers of referrals, wound closure, numbers of wounds and quantity and cost of products used will be collected and compared with the historical record for three months prior to the study. Patients will complete a Quality of Life questionnaire at enrolment and exit from the study.

Patients for whom BSN medical UK products are not appropriate or not desired by the patient will not be enrolled and will receive the usual range of products available to the community nursing team.

ELIGIBILITY:
All healthcare professionals of the Billericay team responsible for dressing changes who are willing to take part in this study and give their written informed consent.

Inclusion Criteria for the patients:

* Patients giving their informed consent and with an open wound being treated by the community nursing team
* All patients whose wounds can be treated with BSN medical UK Product range for wound and leg ulcer management.

Exclusion Criteria for the patients:

* Age <18 years
* Subjects who do not give their consent for any reason
* Subjects who are unable to read and understand patient information sheet and consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Incidence of inappropriate use of dressings for the wound condition and patient lifestyle | At the end of 12 weeks treatment period
  As measured by referrals for case review to the Tissue Viability Team during the study

SECONDARY OUTCOMES:
Number of patients with wounds treated | At the end of 12 weeks treatment period
Wound types treated | At the end of 12 weeks treatment period
Total number of wound closure occurred | At the end of 12 weeks treatment period
Average duration of treatment | At the end of 12 weeks treatment period
Patients Quality of Life living with a Wound | At the start of the study and at the end of 12 weeks treatment period
  as measured by use of the validated questionnaire Wound QoL.
Confidence of healthcare professionals in their dressing selection | At the start of the study and at the end of 12 weeks treatment period
  as measured by written assessment
Visual Analogue Scoring by the healthcare professionals of the simplification of training | At the end of 12 weeks treatment period
Time required for training | At the end of 12 weeks treatment period
NHS Trainer's time | At the end of 12 weeks treatment period
NHS Trainer's cost | At the end of 12 weeks treatment period
Nurse's concordance with training measured by the total number of referrals to the tissue viability team caused by inappropriate dressing selections defined by the trust's guidelines | At the end of 12 weeks treatment period
Costs of dressings used | At the end of 12 weeks treatment period
Number of wounds which could not be treated by the integrated range | At the end of 12 weeks treatment period
Condition of wounds which could not be treated by the integrated range | At the end of 12 weeks treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Ray Norris, Principal Investigator — North East London NHS Foundation Trust
Locations (1):
- South West Essex Community Services, North East London NHS Foundation Trust, Brentwood Community Hospital, Brentwood, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blome C, Baade K, Debus ES, Price P, Augustin M. The "Wound-QoL": a short questionnaire measuring quality of life in patients with chronic wounds based on three established disease-specific instruments. Wound Repair Regen. 2014 Jul-Aug;22(4):504-14. doi: 10.1111/wrr.12193. PMID 24899053
- [Background] British Broadcasting Corporation 10th Sept 2015 www.bbc.co.uk/news/ accessed 6th Oct 2015
- [Background] Cook L (2011) Assessment: exploring competency and current practice.British Journal of Community Nursing Wound care supplement 16. S34-40
- [Background] Dowsett C (2009) Use of TIME to improve community nurses' wound care knowledge and practice.. Wounds UK, Vol 5 No.3
- [Background] Dowsett C, Bielby A, Searle R. Reconciling increasing wound care demands with available resources. J Wound Care. 2014 Nov;23(11):552, 554, 556-8 passim. doi: 10.12968/jowc.2014.23.11.552. PMID 25375403
- [Background] Guest JF, Ayoub N, McIlwraith T, Uchegbu I, Gerrish A, Weidlich D, Vowden K, Vowden P. Health economic burden that wounds impose on the National Health Service in the UK. BMJ Open. 2015 Dec 7;5(12):e009283. doi: 10.1136/bmjopen-2015-009283. PMID 26644123
- [Background] Huynh T, Forget-Falcicchio C. Assessing the primary nurse role in the wound healing process. J Wound Care. 2005 Oct;14(9):407-9. doi: 10.12968/jowc.2005.14.9.26832. PMID 16240619
- [Background] Joy H, Bielby A, Searle R. A collaborative project to enhance efficiency through dressing change practice. J Wound Care. 2015 Jul;24(7):312, 314-7. doi: 10.12968/jowc.2015.24.7.312. PMID 26198553
- [Background] Kerr (2014) How best to record and describe wound exudate Wounds UK Vol 10 No 2
- [Background] McIntosh C, Ousey K (2008) A survey of nurses' and podiatrists' attitudes, skills and knowledge of lower extremity wound care. Wounds UK Vol 4 No 1
- [Background] Office for National Statistics (2011) Topic Guide to Older People.
- [Background] Ousey K. Stephenson J et al (2013) Wound Care in five English NHS Trusts: Results of a Survey. Wounds UK Vol 9 No 4
- [Background] Smith G, Greenwood M, Searle R. Ward nurses' use of wound dressings before and after a bespoke education programme. J Wound Care. 2010 Sep;19(9):396-402. doi: 10.12968/jowc.2010.19.9.78229. PMID 20852568
- [Background] Wicks G (2012) CQUIN Targets; effective dressing selection. Wound Essentials Vol 7 Issue 2 Nov
- [Background] Wong I. Assessing the value of a leg ulcer education programme in Hong Kong. J Wound Care. 2003 Jan;12(1):17-9. doi: 10.12968/jowc.2003.12.1.26459. PMID 12572232